CLINICAL TRIAL: NCT02438319
Title: Automatic vs. Manual Optic Cup and Optic Disc Segmentation in Glaucoma
Brief Title: Automatic vs. Manual Optic Disc Planimetry
Acronym: Planimetry
Status: Withdrawn | Type: Observational
Why Stopped: study was not started
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Optic Disc Planimetry
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with open angle glaucoma: patients with open angle glaucoma who had their optic discs routinely documented by fundus photography. Optic disc photographs will be analyzied by manual planimetry or automated planimetry.
  Interventions: Other: manual planimetry; Other: automated planimetry

INTERVENTIONS:
Other: manual planimetry — Manually marking of the boundaries of the optic disc and it's excavation on color photographs of the optic disc.
Other: automated planimetry — Automatic detection of the boundaries of the optic disc and it's excavation on color photographs of the optic disc.

SUMMARY:
Manually and automatically by mashing learning algorithm optic disc will be evaluated (planimetry).

DETAILED DESCRIPTION:
Cross-Over non-randomized Case-Series. Arm 1 (Manual segmentation): Manually marking of the boundaries of the optic disc and it's excavation on color photographs of the optic disc. Arm 2 (Automated segmentation): Automatic detection of the boundaries of the optic disc and it's excavation. Calculation of cup size, size of excavation, cup-to-disc ratio, and rim area. Comparison of all parameters of both arms and computing of agreement.

ELIGIBILITY:
Inclusion Criteria:

* open-angle glaucoma

Exclusion Criteria:

* no fundus photography of the optic disc performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of open-angle glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
agreement measured by kappa statistics | Baseline visit in the outpatient department
  agreement measured by kappa statistics

SECONDARY OUTCOMES:
Cup size | Baseline visit in the outpatient department
  Cup size
size of excavation | Baseline visit in the outpatient department
  size of excavation
vertical cup to disc ratio | Baseline visit in the outpatient department
  vertical cup to disc ratio
rim area | Baseline visit in the outpatient department
  rim area

CONTACTS AND LOCATIONS:
Overall Officials: Jens Funk, MD, PhD, Principal Investigator — University of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jonas JB. [Glaucoma diagnosis of the optic disc using photography and planimetry]. Ophthalmologe. 2003 Jan;100(1):13-20. doi: 10.1007/s00347-002-0752-4. German. PMID 12557021